CLINICAL TRIAL: NCT03256643
Title: Cognitive and Physical Effects of Exercise or Exercise With Enrichment on People With TBI
Brief Title: Brain Injury Therapy of Exercise and Enriched Environment
Acronym: BITEEE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Jay M Meythaler, Professor of Medicine with Tenure, Wayne State University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 123
Record Dates: First submitted 2014-12-09; First posted 2017-08-22 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Brain Injuries
Keywords: traumatic brain injury; brain contusion; craniocerebral trauma; exercise therapy; chronic brain injury; environment impact; cognitive therapy; health facility environment
MeSH Terms: conditions — Brain Injuries; Brain Injuries, Traumatic; Brain Contusion; Craniocerebral Trauma; Brain Injury, Chronic | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise (Experimental): Exercise is the intervention. People be tested before the start of, and after the end of the eight (8) week exercise program.
  Interventions: Behavioral: Exercise
- Delayed Exercise (Experimental): Delayed Exercise Group will have exercise as intervention. People be tested before the start of, and after the end of the eight (8) weeks then after exercise intervention.
  Interventions: Behavioral: Delayed Exercise
- Exercise and Enrichment (Experimental): Exercise and Enrichment Group is the intervention. The group will be tested at the beginning and end of their exercise/enrichment program.
  Interventions: Behavioral: Exercise and enrichment

INTERVENTIONS:
Behavioral: Exercise — Exercise intervention will consist of 8 exercise classes and exercises at home. A booklet will be given to each person that has a description and photograph of each exercise that designed to work on core strength and balance.
  Arms: Exercise
Behavioral: Delayed Exercise — People will be tested up to 40 weeks after beginning the intervention.
  Arms: Delayed Exercise
Behavioral: Exercise and enrichment — Exercise and enrichment will consist of the same exercise program described for the exercise intervention. The enrichment protocol consisting of cultural educational program will take place during the exercises and breaks for this group.
  Arms: Exercise and Enrichment

SUMMARY:
The purpose of this study is to determine whether exercise or exercise with enrichment is beneficial in individuals who previously had a head injury. The enrichment will consist of a cultural educational program that will include ethnic food, music, slides and a talk. A series of tests that measure mental function and balance will be done before and after the exercise or the exercise/enrichment program will be done to measure efficacy.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) results in long-lasting physical and cognitive deficits. The purpose of this study is to determine whether exercise or exercise with enrichment is beneficial in individuals who previously had a head injury. The environmental enrichment will consist of a cultural educational program that will include ethnic food, music, slides and a talk on 8 different cultures. Individuals will be evaluated using neuropsychological and physical tests before and after the intervention. Testing will consist of Repeatable Battery for the Assessment of Neuropsychological Status (RBANS), Trailmaking Test (TMT), Immediate Post-Concussion Assessment and Cognitive Testing (ImPACT), Quality of Life in Brain Injury Questionnaire (QOLIBRI), 10 meter walk, and the NIH Toolbox Standing Balance Test. Initial testing will include the Disability Rating Scale to help balance groups (after random assignment) in terms of baseline ability.

In rodents, exercise or an enriched environment after TBI improve cognitive function and motor function and the combination results in even greater improvement. The mechanism of cognitive improvement from exercise or environmental enrichment relates to increases in brain derived neurotrophic factor and neurogenesis in the hippocampus. An additional possible mechanism of the positive effects of exercise or enrichment is a reduction in inflammation. Our hypothesis is that exercise or exercise with enrichment will result in better motor performance and improved cognitive ability.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic brain injury (TBI) person
* 1 to 15 year post-TBI
* Initial Glascow Coma SCale (GCS) of < or = 12
* 18-75 years old
* able to perform standardized exercise program

Exclusion Criteria

* Inability to walk independently without assistive aids.
* Severe cardiovascular limitations limiting exercise of up to 5 metabolic equivalents.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Trail Making Part B | Change from Baseline at 9 weeks.
  Trail Making test is a measure of visual conceptual and visuomotor tracking, attention, and maintenance of cognitive set-shifting that is known to be highly sensitive to brain damage.

SECONDARY OUTCOMES:
Quality of Life in Brain Injury Questionnaire | Change from Baseline at 9 weeks.
  Quality of Life in Brain Injury Questionnaire is a thirty-seven question self-reported measure of overall patient health.

OTHER OUTCOMES:
Immediate Post-Concussion Assessment and Cognitive Testing (ImPACT) | Change from Baseline at 9 weeks.
  ImPACT is a measure which consists of a word discrimination, design memory, X/O, symbol matching, color matching, and three letter memory tasks.
Ten Minute Walk | Change from Baseline at 9 weeks.
  Ten Meter Walk is a physical measure of balance and gait, consisting of measuring the time it takes for participants to walk.
NIH Toolbox Standing Balance Test | Change from Baseline and at 9 weeks.
  Standing Balance Test measures the detection of spatial orientation, maintenance of posture in static and dynamic conditions.
Repeatable Battery for the Assessment of Neuropsychological Status | Change from Baseline at 9 weeks.
  is a measure of immediate memory, visuospatial/constructional skills, language, attention, and delayed memory.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Peduzzi-Nelson, Ph.D., Study Director — Wayne State University I
Locations (1):
- Oakwood Heritage, Taylor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alwis DS, Rajan R. Environmental enrichment and the sensory brain: the role of enrichment in remediating brain injury. Front Syst Neurosci. 2014 Sep 2;8:156. doi: 10.3389/fnsys.2014.00156. eCollection 2014. PMID 25228861
- [Background] Bondi CO, Klitsch KC, Leary JB, Kline AE. Environmental enrichment as a viable neurorehabilitation strategy for experimental traumatic brain injury. J Neurotrauma. 2014 May 15;31(10):873-88. doi: 10.1089/neu.2014.3328. Epub 2014 Apr 17. PMID 24555571
- [Background] Fischer FR, Peduzzi JD. Functional recovery in rats with chronic spinal cord injuries after exposure to an enriched environment. J Spinal Cord Med. 2007;30(2):147-55. doi: 10.1080/10790268.2007.11753926. PMID 17591227
- [Background] Gomez-Pinilla F, Hillman C. The influence of exercise on cognitive abilities. Compr Physiol. 2013 Jan;3(1):403-28. doi: 10.1002/cphy.c110063. PMID 23720292
- [Background] Piao CS, Stoica BA, Wu J, Sabirzhanov B, Zhao Z, Cabatbat R, Loane DJ, Faden AI. Late exercise reduces neuroinflammation and cognitive dysfunction after traumatic brain injury. Neurobiol Dis. 2013 Jun;54:252-63. doi: 10.1016/j.nbd.2012.12.017. Epub 2013 Jan 8. PMID 23313314